CLINICAL TRIAL: NCT04784728
Title: A Phase 1, Open Label, Randomized, Three-treatment, Three-sequence, Three-period, Crossover Adhesion Performance and Pharmacokinetic Study of Lidocaine Topical System 1.8% in Healthy, Adult Subjects Under Normal and Two Water Stress Conditions
Brief Title: Pharmacokinetics and Adhesion of Lidocaine Topical System 1.8% With Water Exposure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCI-LIDO-ADH-004
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lidocaine topical system with swimming (Treatment A) (Experimental): One topical system is applied to the mid- to upper-back for 12 hours. Subjects swim for 15 minutes in a heated pool 4 hours after topical system application.
  Interventions: Drug: Lidocaine topical system 1.8%
- Lidocaine topical system with showering (Treatment B) (Experimental): One topical system is applied to the mid- to upper-back for 12 hours. Subjects take a 10-minute shower 8 hours after topical system application.
  Interventions: Drug: Lidocaine topical system 1.8%
- Lidocaine topical system under normal conditions (Treatment C) (Experimental): One topical system is applied to the mid- to upper-back for 12 hours. Topical systems are not exposed to water during this period.
  Interventions: Drug: Lidocaine topical system 1.8%

INTERVENTIONS:
Drug: Lidocaine topical system 1.8% — lidocaine patch
  Other Names: ZTlido

SUMMARY:
The objectives of this study are to evaluate the adhesion performance and pharmacokinetics of ZTlido (lidocaine topical system) 1.8% during swimming, showering, and under normal conditions.

DETAILED DESCRIPTION:
In this Phase 1, open-label, three-period crossover study, 24 healthy, adult male and female subjects are randomized to 1 of 3 treatment sequences. During each treatment period, subjects have one lidocaine topical system applied to their back for 12 hours with a 4-day washout between treatments. In each treatment period, the subject will either swim (Treatment A), shower (Treatment B), or refrain from these activities (Treatment C) while wearing the topical system. Blood samples for lidocaine PK will be collected pre-dose until 24 hours. Adhesion will be monitored throughout the wear time and skin irritation will be assessed the topical system is removed.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy based on medical history, laboratory work, and physical exam
* Body mass index ranging between 18.0-30.0 kg/m2, inclusive
* Capable of unaided swimming
* If childbearing potential, use of acceptable form of birth control
* In case of females of childbearing potential, have a negative serum pregnancy

Key Exclusion Criteria:

* Allergy or known hypersensitivity to lidocaine, amide-type local anesthetics or any component of the product formulation
* Any major medical illness 3 months prior or any significant history or ongoing chronic medical illness affecting the major body systems, including the skin
* Subjects with conditions that might affect application of the product or its adhesive properties (including psoriasis, eczema, atopic dermatitis, damaged or irritated epidermal layer, and excessive hair or oil on the skin)
* Use of antiarrhymthic drugs (such as tocainide and mexiletine) and local anesthetics within 14 days prior to product application.
* History of addiction, abuse, or misuse of any drug
* Use of nicotine-containing products within 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Mean cumulative adhesion score | Over 12 hours
  Adhesion to skin assessed by FDA 0-4 scoring system. The scoring for adhesion of patches is indicated as follows: 0 = ≥ 90% Adhered (essentially no lift off the skin), 1 = ≥ 75% to < 90% Adhered (some edges only lifting off the skin), 2 = ≥ 50% to < 75% Adhered (less than half of the patch lifting off the skin), > 0% to < 50% Adhered but not detached (more than half of the patch lifting off the skin without falling off), and 4 = 0% adhered (patched completely detached). The cumulative adhesion score is calculated as the sum of scores at each assessment time point (3, 4.5, 7, 8.5, and 12 hours).

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of lidocaine | 0, 1.5, 3.0, 6.0, 9.0, 12.0, 15.0, 18.0, 24.0 hours post-dose
  Peak plasma concentration of lidocaine after product application for 12 hours
Area under the plasma concentration-time curve (AUC) from Time 0 to Time 24 hours | 0, 1.5, 3.0, 6.0, 9.0, 12.0, 15.0, 18.0, 24.0 hours post-dose
  Area under the plasma concentration versus time curve from 0 to 24 hours of lidocaine in plasma
Area under the plasma concentration-time curve (AUC) from Time 0 to Time Infinity | 0, 1.5, 3.0, 6.0, 9.0, 12.0, 15.0, 18.0, 24.0 hours post-dose
  Area under the plasma concentration versus time curve from 0 to infinite time of lidocaine in plasma
Dermal Response Score | 12.5 and 14 hours post-dose
  Product tolerability is assessed by Dermal Response Score. The application site is evaluated 30 minutes and 2 hours after product removal (12.5 and 14 hours post-dose, respectively). Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test (i.e., application) site.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boldingh, PharmD, Principal Investigator — AXIS Clinicals
Locations (1):
- AXIS Clinicals, Dilworth, Minnesota, United States

REFERENCES:
- [Derived] Vought K, Greuber E, Patel K, Argoff C, Lissin D. A Randomized, Crossover, Adhesion Performance and Pharmacokinetic Study of a Lidocaine Topical System Under Conditions of Water Exposure in Healthy Subjects. J Pain Res. 2021 Aug 16;14:2459-2467. doi: 10.2147/JPR.S323789. eCollection 2021. PMID 34429646